CLINICAL TRIAL: NCT03506165
Title: Relationship of Periodontitis to Subclinical Atherosclerosis and Long Term Cardiovascular Risk in Patients With Rheumatoid Arthritis
Brief Title: Relationship of Periodontitis and Cardiovascular Risk in Patients With Rheumatoid Arthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shaimaa Salah, principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17200186
Record Dates: First submitted 2018-03-28; First posted 2018-04-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Rheumatoid Arthritis; Periodontitis
MeSH Terms: conditions — Arthritis, Rheumatoid; Periodontitis | interventions — Periodontal Index

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rheumatoid Arthritis with Periodontitis (Experimental): Rheumatoid Arthritis patients with Periodontitis diagnosed after oral examination then treated with Periodontal treatment
  Interventions: Combination Product: Periodontal treatment
- Rheumatoid without Periodontitis (No Intervention): Rheumatoid Arthritis patients without Periodontitis diagnosed after oral examination with. No interventions

INTERVENTIONS:
Combination Product: Periodontal treatment — oral hygiene instructions, periodontal debridement and removal of other etiologic factors
  Arms: Rheumatoid Arthritis with Periodontitis

SUMMARY:
Rheumatoid arthritis (RA) is one of the most common autoimmune inflammatory arthritis affecting 0.5 to 1% population worldwide characterized by synovitis, increased inflammatory markers and progressive bone and cartilage erosion. RA is associated with an increased cardiovascular morbidity and mortality compared with the general population.

DETAILED DESCRIPTION:
Although inflammation has been shown to contribute substantially to the development of cardiovascular diseases (CVDs) in patients with RA, there is also a high prevalence of traditional CVD-risk factors among these patients.

The elevated risk has been shown to be attributable to combination of both traditional risk factors hypertension, smoking, dyslipidemia and obesity and RA-specific factors rheumatoid factor (RF) positivity, rheumatoid factor (RF) positivity and Disease Activity Score including 28 joints (DAS28).

Periodontitis, a chronic inflammatory disease characterized by loss of the periodontal ligament and alveolar bone, is a major cause of tooth loss.

Periodontal diseases are highly prevalent and can affect up to 90% of the world population with varying degree of disease severity. The prevalence of periodontitis is higher in RA population compared to the healthy individuals.

Studies have reported increased periodontal tissue breakdown in RA patients, certain clinical and pathological similarities exist between both diseases. Pathogenic processes in RA, which is characterized by synovial inflammation and progressive destruction of cartilage and bone, are similar to those in periodontitis.

Periodontitis also has been linked to other diseases known to be associated (higher) with RA as diabetes, CVD, metabolic syndrome, some types of cancer.

Periodontitis is one of the major modifiable risk factor of CVD. Both periodontitis and CVD share common risk factors as smoking, diabetes mellitus, age, socioeconomic status, stress and obesity, which could result in confounding any association between them.

Studies revealed that periodontal treatment improves endothelial function and there was a longitudinal study evaluating the impact of periodontal treatment on c-IMT in people with mild/moderate periodontitis. 6 and 12 months following periodontal treatment, a statistically significant reduction in c-IMT compared to baseline measurements was reported. These associations emphasize the importance of oral health as a common under-recognized factor increasing CV risk.

ELIGIBILITY:
Inclusion Criteria:

* The study participants' will be diagnosed according to 2010 ACR/ EULAR classification criteria of rheumatoid arthritis

Exclusion Criteria:

* Participants with history of CVD event (myocardial infarction, coronary artery disease/reperfusion therapy, stroke, transient ischemic attack) in past or any patient experiencing cardiovascular revascularization surgery or the onset of cerebrovascular disorder within past 6 months or those with serious liver disease or renal disease will be excluded, as well.

Patients with overlap diseases will be excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Framingham risk score Low (<10%), Moderate (11-19%) and high risk (>20). | 30 minute
  Examine if there is association between periodontitis with cardiovascular disease risk in patients with RA

CONTACTS AND LOCATIONS:
Overall Officials: Salah, Principal Investigator — Assiut University
Locations (1):
- Assiut university hospitals, Asyut, Egypt

REFERENCES:
- [Background] Aletaha D, Neogi T, Silman AJ, Funovits J, Felson DT, Bingham CO 3rd, Birnbaum NS, Burmester GR, Bykerk VP, Cohen MD, Combe B, Costenbader KH, Dougados M, Emery P, Ferraccioli G, Hazes JM, Hobbs K, Huizinga TW, Kavanaugh A, Kay J, Kvien TK, Laing T, Mease P, Menard HA, Moreland LW, Naden RL, Pincus T, Smolen JS, Stanislawska-Biernat E, Symmons D, Tak PP, Upchurch KS, Vencovsky J, Wolfe F, Hawker G. 2010 Rheumatoid arthritis classification criteria: an American College of Rheumatology/European League Against Rheumatism collaborative initiative. Arthritis Rheum. 2010 Sep;62(9):2569-81. doi: 10.1002/art.27584. PMID 20872595
- [Background] Gibofsky A. Epidemiology, pathophysiology, and diagnosis of rheumatoid arthritis: A Synopsis. Am J Manag Care. 2014 May;20(7 Suppl):S128-35. PMID 25180621
- [Background] Hayashi H, Satoi K, Sato-Mito N, Kaburagi T, Yoshino H, Higaki M, Nishimoto K, Sato K. Nutritional status in relation to adipokines and oxidative stress is associated with disease activity in patients with rheumatoid arthritis. Nutrition. 2012 Nov-Dec;28(11-12):1109-14. doi: 10.1016/j.nut.2012.02.009. PMID 23044162
- [Background] Solomon DH, Karlson EW, Rimm EB, Cannuscio CC, Mandl LA, Manson JE, Stampfer MJ, Curhan GC. Cardiovascular morbidity and mortality in women diagnosed with rheumatoid arthritis. Circulation. 2003 Mar 11;107(9):1303-7. doi: 10.1161/01.cir.0000054612.26458.b2. PMID 12628952
- [Background] Gonzalez A, Maradit Kremers H, Crowson CS, Ballman KV, Roger VL, Jacobsen SJ, O'Fallon WM, Gabriel SE. Do cardiovascular risk factors confer the same risk for cardiovascular outcomes in rheumatoid arthritis patients as in non-rheumatoid arthritis patients? Ann Rheum Dis. 2008 Jan;67(1):64-9. doi: 10.1136/ard.2006.059980. Epub 2007 May 21. PMID 17517756
- [Background] Kawar N, Gajendrareddy PK, Hart TC, Nouneh R, Maniar N, Alrayyes S. Periodontal disease for the primary care physician. Dis Mon. 2011 Apr;57(4):174-83. doi: 10.1016/j.disamonth.2011.03.003. No abstract available. PMID 21569880
- [Background] de Pablo P, Dietrich T, McAlindon TE. Association of periodontal disease and tooth loss with rheumatoid arthritis in the US population. J Rheumatol. 2008 Jan;35(1):70-6. Epub 2007 Nov 15. PMID 18050377
- [Background] Pischon N, Pischon T, Kroger J, Gulmez E, Kleber BM, Bernimoulin JP, Landau H, Brinkmann PG, Schlattmann P, Zernicke J, Buttgereit F, Detert J. Association among rheumatoid arthritis, oral hygiene, and periodontitis. J Periodontol. 2008 Jun;79(6):979-86. doi: 10.1902/jop.2008.070501. PMID 18533773
- [Background] Liljestrand JM, Paju S, Pietiainen M, Buhlin K, Persson GR, Nieminen MS, Sinisalo J, Mantyla P, Pussinen PJ. Immunologic burden links periodontitis to acute coronary syndrome. Atherosclerosis. 2018 Jan;268:177-184. doi: 10.1016/j.atherosclerosis.2017.12.007. Epub 2017 Dec 6. PMID 29232563
- [Background] AlJehani YA. Risk factors of periodontal disease: review of the literature. Int J Dent. 2014;2014:182513. doi: 10.1155/2014/182513. Epub 2014 May 20. PMID 24963294 (Retraction: PMID 33628249 Int J Dent. 2021 Feb 12;2021:8735071)
- [Background] Piconi S, Trabattoni D, Luraghi C, Perilli E, Borelli M, Pacei M, Rizzardini G, Lattuada A, Bray DH, Catalano M, Sparaco A, Clerici M. Treatment of periodontal disease results in improvements in endothelial dysfunction and reduction of the carotid intima-media thickness. FASEB J. 2009 Apr;23(4):1196-204. doi: 10.1096/fj.08-119578. Epub 2008 Dec 12. PMID 19074511